CLINICAL TRIAL: NCT05743842
Title: TriNav Infusion System for the Evaluation of Fidelity Between 99mTc-MAA and Y90-Microspheres Hepatic Distribution for Dosimetry Treatment Planning
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: TriSalus Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-0769; NCI-2023-01620 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TriSalus™ TriNav™Infusion System (catheter) (Experimental): TriNav Infusion System (TriNav catheter) for the injection of the surrogate/test dose during the planning part of the radioembolization procedure and your actual treatment with the radioactive microspheres match each other better than the standard catheter
  Interventions: Device: TriSalus™ TriNav™Infusion System; Diagnostic Test: Angiogram; Procedure: Y90-radioembolization procedure

INTERVENTIONS:
Device: TriSalus™ TriNav™Infusion System — Given by Infusion
Diagnostic Test: Angiogram — X-ray photograph
Procedure: Y90-radioembolization procedure — procedure

SUMMARY:
To learn if using the TriNav Infusion System (TriNav catheter) for the injection of the surrogate/test dose during the planning part of the radioembolization procedure and your actual treatment with the radioactive microspheres match each other better than the standard catheter.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the percentage of tumors that demonstrate quantitative mean dose concordance (within 20%) using voxel-level quantitative SPECT/CT between 99mTc-MAA treatment planning to post therapy Y90 microspheres with an FDA-cleared Pressure Enabled Drug DeliveryTM (PEDDTM) device.

Secondary Objectives:

To determine the correlation of T:N ratios of all tumors 3cm based on 99mTc-MAA SPECT/CT and Y90 SPECT/CT imaging.

To determine the fidelity and concordance of perfused normal liver uptake and distribution between 99mTc-MAA treatment planning to post therapy Y90 microspheres SPECT/CT.

To assess safety of TriNav catheter in this study population

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, of any race or sex, who have unresectable primary or metastatic tumors of the liver, and who are able to give informed consent.
* Patients must be eligible for Y90-radioembolization treatment, have an ECOG Performance Status score of ≤ 2, with a life expectancy of ≥ 3 months, and must be non-pregnant with an acceptable contraception in premenopausal women.
* At least one lesion ≥ 3.0 cm in shortest dimension
* Negative pregnancy test in premenopausal women

Exclusion Criteria:

* Contraindications to angiography and selective visceral catheterization
* Evidence of potential delivery of greater than 30 Gy absorbed dose to the lungs with a single injection.
* Evidence of any detectable Tc-99m MAA flow to the stomach or duodenum, after application of established angiographic techniques to stop or mitigate such flow (eg, placing catheter distal to gastric vessels)
* Infiltrative tumors
* Target vessel sizes outside of TriNav device prescribed diameter range of 1.5 - 3.5 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Armeen Mahvash, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org